CLINICAL TRIAL: NCT05175820
Title: Working Conditions of Dentists During the New Coronavirus (COVID-19) Era
Brief Title: COVID-19 and Working Conditions of Dentists
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Other Study IDs: 2020/47
Record Dates: First submitted 2021-12-29; First posted 2022-01-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Dentistry
Keywords: COVID-19; awareness; dentistry; pandemic; protective measures
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dentists: * Graduated from the Faculty of Dentistry,
  * Continuing/not continuing dental education (master, doctor, doctorate) after graduation,
  * Working in practice or outpatient clinic, private or public hospital, private polyclinic or public health or university hospital,
  * Dentists who registered in Turkish Dental Association
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Survey questions were sent through the mailing list of the Turkish Dental Association, where all dentists in Turkey are registered
  Other Names: questionnaire

SUMMARY:
The aim of this study is to evaluate the protective measures and awareness of dentists working in Turkey regarding the COVID-19 pandemic.

DETAILED DESCRIPTION:
Within the scope of the study, patient care protocols in public and private health institutions during and after the pandemic, published on the website of the Turkish Dental Association (http://www.tdb.org.tr/) A survey consisting of 35 open-ended and multiple-choice questions was prepared based on the updated directive titled.

The questions directed to dentists in the prepared questionnaire are distributed as follows:

* Demographic information (6 questions),
* Physical conditions of the unit to be served (5 questions),
* Applications for employees (2 questions),
* Applications for appointment and patient admission (4 questions),
* Study procedure and treatment protocols (10 questions),
* Attitudes towards COVID-19 (8 questions) Existing questionnaire questions were examined by 5 dentists for clarity and finalized.

A pilot study was conducted on a group of 20 dentists before the prepared questionnaire started to work. The reliability of the questionnaire was evaluated by retesting this group of 20 people 10 days later. 20 people included in the pilot study were evaluated within the scope of the study.

Survey questions were shared online. According to the data of the Turkish Dental Association, survey questions were sent to the registered dentists in the chambers.

Before the survey questions appear on the screen, individuals will be informed of the privacy policy for data collection and consent to volunteering is asked. If they answered "no" to the survey, the survey was closed automatically. A second reminder email was sent to those who did not respond to the questionnaire four days later. A reminder e-mail was sent to those who did not respond to the questionnaire, six days after the start date.

ELIGIBILITY:
Inclusion Criteria:

* Graduated from a dentistry faculty,
* Continuing or not continuing postgraduate dentistry education (master, specialty, doctorate),
* Working in a practice or outpatient clinic, private or public hospital, private polyclinic or state oral and dental health center or university hospital,
* All dentists registered in dentistry database in Turkey (37 cities)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Undergrafute students who have not graduated from the faculty of dentistry,
  * Dentists who are not registered in the Turkish Dental Association
Sampling Method: Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Infection prevention | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Figen Seymen, Prof., Study Director — Department of Pedodontics, Faculty of Dentistry, Istanbul University; Yelda Kasimoglu Eldem, Assoc. Prof., Principal Investigator — Department of Pedodontics, Faculty of Dentistry, Istanbul University
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No